CLINICAL TRIAL: NCT07297862
Title: Investigation of the Psychometric Properties of the Virtual Reality Sickness Questionnaire in Stroke Patients
Brief Title: Virtual Reality Sickness Questionnaire: Psychometrics in Stroke Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Beyzanur ŞENTÜRK, Research Assistant, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-BS-001
Record Dates: First submitted 2025-11-19; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Motion Sickness
Keywords: Motion Sickness; Virtual Reality Sickness Questionnaire; Psychometric Properties; Stroke
MeSH Terms: conditions — Motion Sickness; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke Group
  Interventions: Other: Roller Coaster application
- Healthy Group
  Interventions: Other: Roller Coaster application

INTERVENTIONS:
Other: Roller Coaster application — Participants will experience a 15-minute roller coaster virtual reality (VR) for three consecutive days, once a day. During this study, the virtual reality application will be performed while sitting in a chair and while fixed to the chair. The practitioner will be present with the participant throughout the VR application.

SUMMARY:
The aim of this study is to examine the effects of virtual reality on physiological factors (heart rate, blood pressure) in stroke patients and the psychometric properties of the Virtual Reality Sickness Questionnaire in assessing Motion Sickness resulting from virtual reality use.

DETAILED DESCRIPTION:
Despite the proven advantages of virtual reality approximately 30% of users report nausea and up to 40% experience eye strain as a result of prolonged exposure to virtual environments and simulators. These problems are referred to as motion sickness (MS) a side effect of virtual reality use.

The Motion Sickness Assessment Questionnaire (MSAQ) and the Simulator Sickness Questionnaire (SSQ), which evaluates the symptoms under four titles (gastrointestinal, central, peripheral and fatigue), are used in the literature to evaluate this effect. However, these questionnaires may not be sufficient to assess the MS symptoms that develop after virtual reality (VR) applications. Because MS symptoms occur differently in VR and simulation systems. For this reason, the Virtual Reality Sickness Questionnaire (VRSQ) was developed by Kim and his colleagues to evaluate the symptoms that occur after virtual reality. The Turkish validity and reliability of the VRSQ, which consists of 9 questions, was also conducted by Cetin and his friends.

The aim of this study to investigate how virtual reality affects physiological factors (heart rate, blood pressure) in stroke patients and to evaluate the psychometric properties of the Virtual Reality Sickness Questionnaire in assessing VR-induced motion sickness.

ELIGIBILITY:
Inclusion criteria for individuals with stroke:

1. Stroke diagnosis,
2. A minimum score of 24 on the Standardised Mini Mental Test (SMMT), 2.18-80 years old,
3. showing symptoms of MS with a minimum score of 10 on the Virtual Reality Sickness Questionnaire
4. Titmus test result of 3552 arc/s
5. Not having neglect syndrome

Exclusion criteria:

1. Not volunteering for the study,
2. Presence of a diagnosis of neurological disease other than stroke,
3. Presence of a history of previous stroke,
4. Complete or partial loss of vision in one eye,
5. Previous use of Virtual Reality
6. Having diseases affecting the vestibular system such as Vertigo, Benign Paroxysmal Vertigo, Meniere's

Inclusion criteria for Healthy Individuals:

1. A minimum score of 24 on the Standardised Mini Mental Test (SMMT), 2.18-80 years old, 3. showing symptoms of MS with a minimum score of 10 on the Virtual Reality Sickness Questionnaire 4. Titmus test result of 3552 arc/s

Exclusion criteria:

1. Not volunteering for the study,
2. Presence of a diagnosis of neurological disease,
3. Complete or partial loss of vision in one eye,
4. Previous use of Virtual Reality
5. Having diseases affecting the vestibular system such as Vertigo, Benign Paroxysmal Vertigo, Meniere's

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This prospective study will be conducted in BAIBU Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation on healthy individuals and individuals with stroke who agree to participate in the study.
  Individuals between the ages of 18-80 will be included in the study. Individuals will be asked to experience VR for 15 minutes and then fill out the Virtual Reality Sickness Questionnaire. Individuals whose score in this questionnaire is not 10 and above will be excluded from the study. Individuals who meet the inclusion criteria will be divided into two groups as healthy and stroke patients after demographic information is obtained.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2026-08-16 (Estimated)

PRIMARY OUTCOMES:
Virtual Reality Sickness Questionnaire | immediately after roller coaster application
  The Virtual Reality Sickness Questionnaire (VRSQ), which consists of 9 items and two main headings: oculomotor discomfort and disorientation, will be used to assess Motion Sickness symptoms. The items will be scored between 0-3. As a result of VRSQ oculomotor, disorientation and total scores will be obtained. Oculomotor and disorientation scores will be calculated by dividing the individual's component score by the total score obtained (as a percentage). Minimum score is 0 and maximum score is 100. Higher scores mean more symptoms.

SECONDARY OUTCOMES:
Titmus Test | Baseline
  Three-dimensional vision of the participants will be evaluated with the Titmus test with special glasses designed for three-dimensional vision called Binocular vision stereoacuity and a brochure held 40 cm away from eye level. The participant will be asked whether they can see the butterfly on the brochure in three dimensions while wearing the glasses as a yes or no question. Participants who answer yes will proceed to the second stage. In the second stage, they will be asked to say which of the nine squares and four circles in each square they see in three dimensions.
National Institutes of Health Stroke Scale (NIHSS) | Baseline
  With the 15-item National Institutes of Health Stroke Scale (NIHSS), patients with stroke; Very Severe: >25 Severe: 15 - 24 Mild to Moderate: 5 - 14 Mild: 1-5 will be used to classify patients. The test will last 10 minutes and items will be scored as 0-2, 0-3 or 0-4. The maximum score to be obtained from the test is 42.
Standardized Mini Mental Test (SMMT) | Baseline
  For the brief and objective measurement of cognitive function, the Standardized Mini Mental Test (SMMT) will be used, which consists of eleven items grouped under five main headings: orientation, recording memory, attention and calculation, recall and language, and takes 10-15 minutes to administer.
  Severe cognitive impairment: 0-17, Mild cognitive impairment: 18-23, No cognitive impairment: 24-30.
The Motion Sensitivity Test (MST) | immediately after roller coaster application
  The Motion Sensitivity Test (MST) assesses movement-induced dizziness through 16 rapid head and body position changes. For each position, participants report the start and end of dizziness, and duration is scored from 1 to 3 based on time. They also rate dizziness intensity from 0 to 5. Duration and intensity scores are summed to obtain a raw score. The MST quotient is calculated by dividing the total symptom scores by 20.48, with 0 indicating no symptoms and 100 indicating severe symptoms in all positions.
Tolerance Period | During application
  The patient's tolerance period, the time until symptoms become apparent, will be recorded
Heart Rate | baseline and immediately after roller coaster application
  Participants' heart rate will be recorded with a device before and after the virtual reality experience
Feeling of discomfort | immediately after roller coaster application
  Discomfort will be calculated by measuring the area marked by the individual from 0 (very comfortable) to 10 (not comfortable at all).
Blood Pressure | baseline and immediately after roller coaster application
  Participants' blood pressure will be recorded with a device before and after the virtual reality experience

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided